CLINICAL TRIAL: NCT01082588
Title: Phase 4 Study of the Effects of Pravastatin on Cholesterol Levels, Inflammation and Cognition in Schizophrenia
Brief Title: Effects of Pravastatin on Cholesterol, Inflammation and Cognition in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Stanley Medical Research Institute (Other); North Suffolk Mental Health Association (Other)
Responsible Party: Principal Investigator, David C. Henderson, Associate Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-P-002524; 09T-1296 (Other Grant/Funding Number: Stanley Medical Research Institute); NCT01363219 (obsolete NCT alias)
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Results first posted 2014-04-28 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-03

CONDITIONS: Schizophrenia; Schizoaffective Disorders; Schizophreniform Disorders
Keywords: schizophrenia; pravastatin; inflammation; cognition; antipsychotics; cholesterol
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Inflammation | interventions — Pravastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pravastatin (Active Comparator): pravastatin 40mg, once a day, shortly after baseline for 12 consecutive weeks
  Interventions: Drug: Pravastatin
- Placebo (Placebo Comparator): placebo, once a day, shortly after baseline for 12 consecutive weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pravastatin — pravastatin 40mg, or placebo, once a day, shortly after baseline for 12 consecutive weeks
  Other Names: pravastatin sodium; Pravachol
  Arms: pravastatin
Drug: Placebo — pravastatin 40mg, or placebo, once a day, shortly after baseline for 12 consecutive weeks
  Arms: Placebo

SUMMARY:
This study involves people with schizophrenia or schizoaffective disorder, who are currently taking antipsychotic medications. Some antipsychotic medications may cause an increase in cholesterol levels, which may lead to inflammation in the body. Inflammation poses a risk in developing heart disease, diabetes and problems with brain function. The purpose of this study is to see if pravastatin can:

* Lower cholesterol
* Decrease inflammation
* Improve cognition in patients with schizophrenia

DETAILED DESCRIPTION:
This study is a 12-week randomized, double-blind, placebo-controlled pilot study of pravastatin 40mg a day, administered for 12 consecutive weeks to subjects with schizophrenia to examine pravastatin's effects on lowering cholesterol levels and inflammatory markers, and improving cognition. The study will be conducted at the Freedom Trail Clinic and will use the Massachusetts General Hospital Clinical Research Center. The innovative approach of using pravastatin to not only decrease cholesterol levels, but to decrease inflammation and improve cognition in patients with schizophrenia is promising and may lead to a different approach to treatment in this population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18-68 years
* Diagnosis of schizophrenia, any subtype, schizoaffective disorder, any subtype or schizophreniform disorder
* Well established compliance with outpatient medications including their antipsychotic medication

Exclusion Criteria:

* Inability to provide informed consent
* Current substance and alcohol abuse
* Significant medical illness, including congestive heart failure, severe cardiovascular disease, renal disease (serum creatinine > 1.5), severe hepatic impairment or active liver disease, anemia (hemoglobin <11.0 gm/dL), history of severe head injury, and not treated muscle disease.
* Psychiatrically unstable
* Women of child bearing potential who are pregnant, breastfeeding, or who are unwilling or unable to use an effective form of birth control during the entire study
* Subjects treated with anti-inflammatory drugs (including daily aspirin and ibuprofen), thiazide diuretics; agents that induce weight loss, and St. John's Wort will be excluded from the study
* Current history of untreated thyroid disease
* Current treatment with insulin
* Subjects being treated with drugs such as: colchicine, azole antifungals (fluconazole, ketoconazole, itraconazole); macrolide antibiotics (clarithromycin, erythromycin); HIV protease inhibitors (ritonavir, indinavir, saquinavir, nelfinavir) that inhibit the CYP 450 3A liver enzyme
* Known hypersensitivity to pravastatin or any of its components

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David C Henderson, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Freedom Trail Clinic, Boston, Massachusetts, United States

REFERENCES:
- [Background] Muller N, Riedel M, Gruber R, Ackenheil M, Schwarz MJ. The immune system and schizophrenia. An integrative view. Ann N Y Acad Sci. 2000;917:456-67. doi: 10.1111/j.1749-6632.2000.tb05410.x. PMID 11268373
- [Background] Maes M, Bocchio Chiavetto L, Bignotti S, Battisa Tura GJ, Pioli R, Boin F, Kenis G, Bosmans E, de Jongh R, Altamura CA. Increased serum interleukin-8 and interleukin-10 in schizophrenic patients resistant to treatment with neuroleptics and the stimulatory effects of clozapine on serum leukemia inhibitory factor receptor. Schizophr Res. 2002 Apr 1;54(3):281-91. doi: 10.1016/s0920-9964(00)00094-3. PMID 11950553
- [Background] Sirota P, Meiman M, Herschko R, Bessler H. Effect of neuroleptic administration on serum levels of soluble IL-2 receptor-alpha and IL-1 receptor antagonist in schizophrenic patients. Psychiatry Res. 2005 Apr 15;134(2):151-9. doi: 10.1016/j.psychres.2004.04.012. PMID 15840416
- [Background] Rapaport MH, Lohr JB. Serum-soluble interleukin-2 receptors in neuroleptic-naive schizophrenic subjects and in medicated schizophrenic subjects with and without tardive dyskinesia. Acta Psychiatr Scand. 1994 Nov;90(5):311-5. doi: 10.1111/j.1600-0447.1994.tb01599.x. PMID 7872033
- [Background] Potvin S, Stip E, Sepehry AA, Gendron A, Bah R, Kouassi E. Inflammatory cytokine alterations in schizophrenia: a systematic quantitative review. Biol Psychiatry. 2008 Apr 15;63(8):801-8. doi: 10.1016/j.biopsych.2007.09.024. Epub 2007 Nov 19. PMID 18005941
- [Background] Naudin J, Capo C, Giusano B, Mege JL, Azorin JM. A differential role for interleukin-6 and tumor necrosis factor-alpha in schizophrenia? Schizophr Res. 1997 Aug 29;26(2-3):227-33. doi: 10.1016/s0920-9964(97)00059-5. PMID 9323355
- [Background] Monteleone P, Fabrazzo M, Tortorella A, Maj M. Plasma levels of interleukin-6 and tumor necrosis factor alpha in chronic schizophrenia: effects of clozapine treatment. Psychiatry Res. 1997 Jun 16;71(1):11-7. doi: 10.1016/s0165-1781(97)00036-x. PMID 9247977
- [Background] Boin F, Zanardini R, Pioli R, Altamura CA, Maes M, Gennarelli M. Association between -G308A tumor necrosis factor alpha gene polymorphism and schizophrenia. Mol Psychiatry. 2001 Jan;6(1):79-82. doi: 10.1038/sj.mp.4000815. PMID 11244489
- [Background] Meira-Lima IV, Pereira AC, Mota GF, Floriano M, Araujo F, Mansur AJ, Krieger JE, Vallada H. Analysis of a polymorphism in the promoter region of the tumor necrosis factor alpha gene in schizophrenia and bipolar disorder: further support for an association with schizophrenia. Mol Psychiatry. 2003 Aug;8(8):718-20. doi: 10.1038/sj.mp.4001309. No abstract available. PMID 12888800
- [Background] Bouma G, Crusius JB, Oudkerk Pool M, Kolkman JJ, von Blomberg BM, Kostense PJ, Giphart MJ, Schreuder GM, Meuwissen SG, Pena AS. Secretion of tumour necrosis factor alpha and lymphotoxin alpha in relation to polymorphisms in the TNF genes and HLA-DR alleles. Relevance for inflammatory bowel disease. Scand J Immunol. 1996 Apr;43(4):456-63. doi: 10.1046/j.1365-3083.1996.d01-65.x. PMID 8668926
- [Background] Wilson AG, Symons JA, McDowell TL, McDevitt HO, Duff GW. Effects of a polymorphism in the human tumor necrosis factor alpha promoter on transcriptional activation. Proc Natl Acad Sci U S A. 1997 Apr 1;94(7):3195-9. doi: 10.1073/pnas.94.7.3195. PMID 9096369
- [Background] McAllister CG, van Kammen DP, Rehn TJ, Miller AL, Gurklis J, Kelley ME, Yao J, Peters JL. Increases in CSF levels of interleukin-2 in schizophrenia: effects of recurrence of psychosis and medication status. Am J Psychiatry. 1995 Sep;152(9):1291-7. doi: 10.1176/ajp.152.9.1291. PMID 7653683
- [Background] Zhang XY, Zhou DF, Cao LY, Zhang PY, Wu GY, Shen YC. Changes in serum interleukin-2, -6, and -8 levels before and during treatment with risperidone and haloperidol: relationship to outcome in schizophrenia. J Clin Psychiatry. 2004 Jul;65(7):940-7. doi: 10.4088/jcp.v65n0710. PMID 15291683
- [Background] Fan X, Pristach C, Liu EY, Freudenreich O, Henderson DC, Goff DC. Elevated serum levels of C-reactive protein are associated with more severe psychopathology in a subgroup of patients with schizophrenia. Psychiatry Res. 2007 Jan 15;149(1-3):267-71. doi: 10.1016/j.psychres.2006.07.011. Epub 2006 Nov 16. PMID 17112596
- [Background] Muller N, Riedel M, Scheppach C, Brandstatter B, Sokullu S, Krampe K, Ulmschneider M, Engel RR, Moller HJ, Schwarz MJ. Beneficial antipsychotic effects of celecoxib add-on therapy compared to risperidone alone in schizophrenia. Am J Psychiatry. 2002 Jun;159(6):1029-34. doi: 10.1176/appi.ajp.159.6.1029. PMID 12042193
- [Background] Rapaport MH, Delrahim KK, Bresee CJ, Maddux RE, Ahmadpour O, Dolnak D. Celecoxib augmentation of continuously ill patients with schizophrenia. Biol Psychiatry. 2005 Jun 15;57(12):1594-6. doi: 10.1016/j.biopsych.2005.02.024. PMID 15953498
- [Background] Dziedzic T. Systemic inflammatory markers and risk of dementia. Am J Alzheimers Dis Other Demen. 2006 Aug-Sep;21(4):258-62. doi: 10.1177/1533317506289260. PMID 16948290
- [Background] Licastro F, Pedrini S, Caputo L, Annoni G, Davis LJ, Ferri C, Casadei V, Grimaldi LM. Increased plasma levels of interleukin-1, interleukin-6 and alpha-1-antichymotrypsin in patients with Alzheimer's disease: peripheral inflammation or signals from the brain? J Neuroimmunol. 2000 Feb 1;103(1):97-102. doi: 10.1016/s0165-5728(99)00226-x. PMID 10674995
- [Background] Bruunsgaard H, Andersen-Ranberg K, Jeune B, Pedersen AN, Skinhoj P, Pedersen BK. A high plasma concentration of TNF-alpha is associated with dementia in centenarians. J Gerontol A Biol Sci Med Sci. 1999 Jul;54(7):M357-64. doi: 10.1093/gerona/54.7.m357. PMID 10462168
- [Background] Yaffe K, Lindquist K, Penninx BW, Simonsick EM, Pahor M, Kritchevsky S, Launer L, Kuller L, Rubin S, Harris T. Inflammatory markers and cognition in well-functioning African-American and white elders. Neurology. 2003 Jul 8;61(1):76-80. doi: 10.1212/01.wnl.0000073620.42047.d7. PMID 12847160
- [Background] Tan ZS, Beiser AS, Vasan RS, Roubenoff R, Dinarello CA, Harris TB, Benjamin EJ, Au R, Kiel DP, Wolf PA, Seshadri S. Inflammatory markers and the risk of Alzheimer disease: the Framingham Study. Neurology. 2007 May 29;68(22):1902-8. doi: 10.1212/01.wnl.0000263217.36439.da. PMID 17536046
- [Background] Etminan M, Gill S, Samii A. Effect of non-steroidal anti-inflammatory drugs on risk of Alzheimer's disease: systematic review and meta-analysis of observational studies. BMJ. 2003 Jul 19;327(7407):128. doi: 10.1136/bmj.327.7407.128. PMID 12869452
- [Background] Dickerson F, Stallings C, Origoni A, Boronow J, Yolken R. C-reactive protein is associated with the severity of cognitive impairment but not of psychiatric symptoms in individuals with schizophrenia. Schizophr Res. 2007 Jul;93(1-3):261-5. doi: 10.1016/j.schres.2007.03.022. Epub 2007 May 8. PMID 17490859
- [Background] Meyer JM, McEvoy JP, Davis VG, Goff DC, Nasrallah HA, Davis SM, Hsiao JK, Swartz MS, Stroup TS, Lieberman JA. Inflammatory markers in schizophrenia: comparing antipsychotic effects in phase 1 of the clinical antipsychotic trials of intervention effectiveness study. Biol Psychiatry. 2009 Dec 1;66(11):1013-22. doi: 10.1016/j.biopsych.2009.06.005. Epub 2009 Jul 29. PMID 19640511
- [Background] Fenton WS, Hibbeln J, Knable M. Essential fatty acids, lipid membrane abnormalities, and the diagnosis and treatment of schizophrenia. Biol Psychiatry. 2000 Jan 1;47(1):8-21. doi: 10.1016/s0006-3223(99)00092-x. PMID 10650444
- [Background] Tracey KJ. The inflammatory reflex. Nature. 2002 Dec 19-26;420(6917):853-9. doi: 10.1038/nature01321. PMID 12490958
- [Background] Laflamme N, Rivest S. Effects of systemic immunogenic insults and circulating proinflammatory cytokines on the transcription of the inhibitory factor kappaB alpha within specific cellular populations of the rat brain. J Neurochem. 1999 Jul;73(1):309-21. doi: 10.1046/j.1471-4159.1999.0730309.x. PMID 10386984
- [Background] Ek M, Engblom D, Saha S, Blomqvist A, Jakobsson PJ, Ericsson-Dahlstrand A. Inflammatory response: pathway across the blood-brain barrier. Nature. 2001 Mar 22;410(6827):430-1. doi: 10.1038/35068632. No abstract available. PMID 11260702
- [Background] Perry VH, Cunningham C, Holmes C. Systemic infections and inflammation affect chronic neurodegeneration. Nat Rev Immunol. 2007 Feb;7(2):161-7. doi: 10.1038/nri2015. Epub 2007 Jan 15. PMID 17220915
- [Background] Sjoholm A, Nystrom T. Inflammation and the etiology of type 2 diabetes. Diabetes Metab Res Rev. 2006 Jan-Feb;22(1):4-10. doi: 10.1002/dmrr.568. PMID 15991254
- [Background] Hotamisligil GS, Shargill NS, Spiegelman BM. Adipose expression of tumor necrosis factor-alpha: direct role in obesity-linked insulin resistance. Science. 1993 Jan 1;259(5091):87-91. doi: 10.1126/science.7678183.
- [Background] Dandona P, Aljada A, Chaudhuri A, Mohanty P. Endothelial dysfunction, inflammation and diabetes. Rev Endocr Metab Disord. 2004 Aug;5(3):189-97. doi: 10.1023/B:REMD.0000032407.88070.0a. No abstract available. PMID 15211090
- [Background] Hotamisligil GS, Peraldi P, Budavari A, Ellis R, White MF, Spiegelman BM. IRS-1-mediated inhibition of insulin receptor tyrosine kinase activity in TNF-alpha- and obesity-induced insulin resistance. Science. 1996 Feb 2;271(5249):665-8. doi: 10.1126/science.271.5249.665. PMID 8571133
- [Background] McEvoy JP, Meyer JM, Goff DC, Nasrallah HA, Davis SM, Sullivan L, Meltzer HY, Hsiao J, Scott Stroup T, Lieberman JA. Prevalence of the metabolic syndrome in patients with schizophrenia: baseline results from the Clinical Antipsychotic Trials of Intervention Effectiveness (CATIE) schizophrenia trial and comparison with national estimates from NHANES III. Schizophr Res. 2005 Dec 1;80(1):19-32. doi: 10.1016/j.schres.2005.07.014. Epub 2005 Aug 30. PMID 16137860
- [Background] Ford DE, Erlinger TP. Depression and C-reactive protein in US adults: data from the Third National Health and Nutrition Examination Survey. Arch Intern Med. 2004 May 10;164(9):1010-4. doi: 10.1001/archinte.164.9.1010. PMID 15136311
- [Background] Lakka HM, Laaksonen DE, Lakka TA, Niskanen LK, Kumpusalo E, Tuomilehto J, Salonen JT. The metabolic syndrome and total and cardiovascular disease mortality in middle-aged men. JAMA. 2002 Dec 4;288(21):2709-16. doi: 10.1001/jama.288.21.2709. PMID 12460094
- [Background] Newcomer JW, Haupt DW, Fucetola R, Melson AK, Schweiger JA, Cooper BP, Selke G. Abnormalities in glucose regulation during antipsychotic treatment of schizophrenia. Arch Gen Psychiatry. 2002 Apr;59(4):337-45. doi: 10.1001/archpsyc.59.4.337. PMID 11926934
- [Background] Henderson DC, Cagliero E, Copeland PM, Borba CP, Evins AE, Hayden D, Weber MT, Anderson EJ, Allison DB, Daley TB, Schoenfeld D, Goff DC. Glucose metabolism in patients with schizophrenia treated with atypical antipsychotic agents: a frequently sampled intravenous glucose tolerance test and minimal model analysis. Arch Gen Psychiatry. 2005 Jan;62(1):19-28. doi: 10.1001/archpsyc.62.1.19. PMID 15630069
- [Background] Bonora E, Kiechl S, Willeit J, Oberhollenzer F, Egger G, Targher G, Alberiche M, Bonadonna RC, Muggeo M. Prevalence of insulin resistance in metabolic disorders: the Bruneck Study. Diabetes. 1998 Oct;47(10):1643-9. doi: 10.2337/diabetes.47.10.1643. PMID 9753305
- [Background] Kitabchi AE, Temprosa M, Knowler WC, Kahn SE, Fowler SE, Haffner SM, Andres R, Saudek C, Edelstein SL, Arakaki R, Murphy MB, Shamoon H; Diabetes Prevention Program Research Group. Role of insulin secretion and sensitivity in the evolution of type 2 diabetes in the diabetes prevention program: effects of lifestyle intervention and metformin. Diabetes. 2005 Aug;54(8):2404-14. doi: 10.2337/diabetes.54.8.2404. PMID 16046308
- [Background] Lillioja S, Mott DM, Spraul M, Ferraro R, Foley JE, Ravussin E, Knowler WC, Bennett PH, Bogardus C. Insulin resistance and insulin secretory dysfunction as precursors of non-insulin-dependent diabetes mellitus. Prospective studies of Pima Indians. N Engl J Med. 1993 Dec 30;329(27):1988-92. doi: 10.1056/NEJM199312303292703. PMID 8247074
- [Background] Semenkovich CF. Insulin resistance and atherosclerosis. J Clin Invest. 2006 Jul;116(7):1813-22. doi: 10.1172/JCI29024. PMID 16823479
- [Background] Weyer C, Tataranni PA, Bogardus C, Pratley RE. Insulin resistance and insulin secretory dysfunction are independent predictors of worsening of glucose tolerance during each stage of type 2 diabetes development. Diabetes Care. 2001 Jan;24(1):89-94. doi: 10.2337/diacare.24.1.89. PMID 11194248
- [Background] Wellen KE, Hotamisligil GS. Inflammation, stress, and diabetes. J Clin Invest. 2005 May;115(5):1111-9. doi: 10.1172/JCI25102. PMID 15864338
- [Background] Nissen SE. Does intensive statin therapy lower mortality and cardiovascular event risk in patients with acute coronary syndrome? Nat Clin Pract Cardiovasc Med. 2005 Jan;2(1):10-1. doi: 10.1038/ncpcardio0066. No abstract available. PMID 16265333
- [Background] Nissen SE, Tuzcu EM, Schoenhagen P, Crowe T, Sasiela WJ, Tsai J, Orazem J, Magorien RD, O'Shaughnessy C, Ganz P; Reversal of Atherosclerosis with Aggressive Lipid Lowering (REVERSAL) Investigators. Statin therapy, LDL cholesterol, C-reactive protein, and coronary artery disease. N Engl J Med. 2005 Jan 6;352(1):29-38. doi: 10.1056/NEJMoa042000. PMID 15635110
- [Background] Ridker PM, Morrow DA, Rose LM, Rifai N, Cannon CP, Braunwald E. Relative efficacy of atorvastatin 80 mg and pravastatin 40 mg in achieving the dual goals of low-density lipoprotein cholesterol <70 mg/dl and C-reactive protein <2 mg/l: an analysis of the PROVE-IT TIMI-22 trial. J Am Coll Cardiol. 2005 May 17;45(10):1644-8. doi: 10.1016/j.jacc.2005.02.080. Epub 2005 Apr 25. PMID 15893181
- [Background] Kaesemeyer WH, Caldwell RB, Huang J, Caldwell RW. Pravastatin sodium activates endothelial nitric oxide synthase independent of its cholesterol-lowering actions. J Am Coll Cardiol. 1999 Jan;33(1):234-41. doi: 10.1016/s0735-1097(98)00514-2. PMID 9935036
- [Background] Harris JI, Hibbeln JR, Mackey RH, Muldoon MF. Statin treatment alters serum n-3 and n-6 fatty acids in hypercholesterolemic patients. Prostaglandins Leukot Essent Fatty Acids. 2004 Oct;71(4):263-9. doi: 10.1016/j.plefa.2004.06.001. PMID 15310527
- [Background] Agrawal A. CRP after 2004. Mol Immunol. 2005 May;42(8):927-30. doi: 10.1016/j.molimm.2004.09.028. Epub 2004 Dec 7. PMID 15829284
- [Background] Black S, Kushner I, Samols D. C-reactive Protein. J Biol Chem. 2004 Nov 19;279(47):48487-90. doi: 10.1074/jbc.R400025200. Epub 2004 Aug 26. PMID 15337754
- [Background] Ridker PM, Cannon CP, Morrow D, Rifai N, Rose LM, McCabe CH, Pfeffer MA, Braunwald E; Pravastatin or Atorvastatin Evaluation and Infection Therapy-Thrombolysis in Myocardial Infarction 22 (PROVE IT-TIMI 22) Investigators. C-reactive protein levels and outcomes after statin therapy. N Engl J Med. 2005 Jan 6;352(1):20-8. doi: 10.1056/NEJMoa042378. PMID 15635109
- [Background] Vuletic S, Riekse RG, Marcovina SM, Peskind ER, Hazzard WR, Albers JJ. Statins of different brain penetrability differentially affect CSF PLTP activity. Dement Geriatr Cogn Disord. 2006;22(5-6):392-8. doi: 10.1159/000095679. Epub 2006 Sep 7. PMID 16960448
- [Background] Ventura J, Liberman RP, Green MF, Shaner A, Mintz J. Training and quality assurance with the Structured Clinical Interview for DSM-IV (SCID-I/P). Psychiatry Res. 1998 Jun 15;79(2):163-73. doi: 10.1016/s0165-1781(98)00038-9. PMID 9705054
- [Background] Kay SR, Opler LA, Lindenmayer JP. The Positive and Negative Syndrome Scale (PANSS): rationale and standardisation. Br J Psychiatry Suppl. 1989 Nov;(7):59-67. No abstract available. PMID 2619982
- [Background] Rey JM, Hunt GE, Johnson GF. Assessment of tardive dyskinesia in psychiatric outpatients using a standardized rating scale. Aust N Z J Psychiatry. 1981 Mar;15(1):33-7. doi: 10.3109/00048678109159407. PMID 6973337
- [Background] HAMILTON M. A rating scale for depression. J Neurol Neurosurg Psychiatry. 1960 Feb;23(1):56-62. doi: 10.1136/jnnp.23.1.56. No abstract available. PMID 14399272
- [Background] Heinrichs DW, Hanlon TE, Carpenter WT Jr. The Quality of Life Scale: an instrument for rating the schizophrenic deficit syndrome. Schizophr Bull. 1984;10(3):388-98. doi: 10.1093/schbul/10.3.388. PMID 6474101
- [Background] Endicott J, Spitzer RL, Fleiss JL, Cohen J. The global assessment scale. A procedure for measuring overall severity of psychiatric disturbance. Arch Gen Psychiatry. 1976 Jun;33(6):766-71. doi: 10.1001/archpsyc.1976.01770060086012. PMID 938196
- [Background] Nuechterlein KH, Green MF, Kern RS, Baade LE, Barch DM, Cohen JD, Essock S, Fenton WS, Frese FJ 3rd, Gold JM, Goldberg T, Heaton RK, Keefe RS, Kraemer H, Mesholam-Gately R, Seidman LJ, Stover E, Weinberger DR, Young AS, Zalcman S, Marder SR. The MATRICS Consensus Cognitive Battery, part 1: test selection, reliability, and validity. Am J Psychiatry. 2008 Feb;165(2):203-13. doi: 10.1176/appi.ajp.2007.07010042. Epub 2008 Jan 2. PMID 18172019
- [Background] Kern RS, Nuechterlein KH, Green MF, Baade LE, Fenton WS, Gold JM, Keefe RS, Mesholam-Gately R, Mintz J, Seidman LJ, Stover E, Marder SR. The MATRICS Consensus Cognitive Battery, part 2: co-norming and standardization. Am J Psychiatry. 2008 Feb;165(2):214-20. doi: 10.1176/appi.ajp.2007.07010043. Epub 2008 Jan 2. PMID 18172018
- [Background] Patterson TL, Goldman S, McKibbin CL, Hughs T, Jeste DV. UCSD Performance-Based Skills Assessment: development of a new measure of everyday functioning for severely mentally ill adults. Schizophr Bull. 2001;27(2):235-45. doi: 10.1093/oxfordjournals.schbul.a006870. PMID 11354591
- [Background] Schakel SF, Sievert YA, Buzzard IM. Sources of data for developing and maintaining a nutrient database. J Am Diet Assoc. 1988 Oct;88(10):1268-71. PMID 3171020
- [Background] McNamara JR, Schaefer EJ. Automated enzymatic standardized lipid analyses for plasma and lipoprotein fractions. Clin Chim Acta. 1987 Jun 30;166(1):1-8. doi: 10.1016/0009-8981(87)90188-4. PMID 3608193
- [Background] Warnick GR, Benderson J, Albers JJ. Dextran sulfate-Mg2+ precipitation procedure for quantitation of high-density-lipoprotein cholesterol. Clin Chem. 1982 Jun;28(6):1379-88. No abstract available. PMID 7074948
- [Background] Friedewald WT, Levy RI, Fredrickson DS. Estimation of the concentration of low-density lipoprotein cholesterol in plasma, without use of the preparative ultracentrifuge. Clin Chem. 1972 Jun;18(6):499-502. No abstract available. PMID 4337382
- [Background] Otvos JD. Measurement of lipoprotein subclass profiles by nuclear magnetic resonance spectroscopy. Clin Lab. 2002;48(3-4):171-80. No abstract available. PMID 11934219
- [Background] Levine S. The management of resistant depression. Acta Psychiatr Belg. 1986 Mar-Apr;86(2):141-51. PMID 3088916

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited from the Massachusetts General Hospital Schizophrenia Clinical and Research Program.
Period: Overall Study
Arm/Group | Pravastatin | Placebo
Started | 30 | 30
Completed | 24 | 25
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pravastatin | Placebo | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.11 (11.06) | 45.08 (12.54) | 44.84 (11.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 14 | 22
  Male | 22 | 16 | 38
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in LDL-cholesterol Between Baseline and Week 12
Time Frame: Baseline, week 12
Population: One participant from the pravastatin group and two from the placebo group had triglyceride levels above 400. Per Massachusetts General Hospital Laboratories policy, LDL is not run as a part of the complete metabolic panel (CMP) when triglycerides are above 400, and therefore could not be included in the final analysis.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 23 | 23
mg/dl | -25.565 (32.261) | -2.913 (16.434)

2. Primary Outcome: Change in C-Reactive Protein (CRP) From Baseline to Week 12
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 24 | 25
mg/L | 0.8063 (5.3515) | -0.5136 (7.2646)

3. Primary Outcome: Change in MATRICS Neuropsychological Battery Composite Score From Baseline to Week 12
Description: The Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery measures cognitive functioning within 7 domains: speed of processing, attention/vigilance, working memory (non verbal and verbal), verbal learning, visual learning, reasoning and problem solving and social cognition.
  The composite score is calculated by the MATRICS computer program, which equally weights each of the 7 domain scores. The range of composite scores is 20-80. Higher scores indicate higher levels or cognitive functioning, while lower scores indicate lower levels of cognitive functioning.
Time Frame: Baseline, week 12
Population: One participant from the placebo group refused to complete the MATRICS assessment at week 12; therefore, we could only analyze 24 placebo participants for the final analysis.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 24 | 24
Scores on a scale | 4.0417 (5.2789) | 4.125 (6.9739)

4. Primary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) Total Score From Baseline to Week 12
Description: The Positive and Negative Syndrome Scale (PANSS) is a scale used to rate severity of schizophrenia. All items are summed to calculate the total score. The scale range is 30-210. Better outcomes have lower numbers and worse outcomes have higher numbers.
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 24 | 25
Scores on a scale | -9.416 (13.941) | -6.48 (12.003)

5. Primary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) Positive Score From Baseline to Week 12
Description: This is a subscale of the Positive and Negative Syndrome Scale (PANSS). The range for this subscale is 7-49. All items are summed to calculate the total score. Better outcomes have lower numbers and worse outcomes have higher numbers.
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 24 | 25
Scores on a scale | -2.9583 (3.014) | -2.44 (4.164)

6. Primary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) Negative Score From Baseline to Week 12
Description: as for outcome 5
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 24 | 25
Scores on a scale | -0.83 (5.411) | -0.28 (3.736)

7. Primary Outcome: Change in Positive and Negative Syndrome Scale (PANSS) General Score From Baseline to Week 12
Description: This is a subscale of the Positive and Negative Syndrome Scale (PANSS). The range for this subscale is 15-105. All items are summed to calculate the total score. Better outcomes have lower numbers and worse outcomes have higher numbers.
Time Frame: Baseline, week 12
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Pravastatin | Placebo
Number analyzed (Participants) | 24 | 25
Scores on a scale | -5.625 (8.155) | -3.76 (6.418)

ADVERSE EVENTS:
Arm/Group | Pravastatin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 5/30 | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pravastatin (N=30) | Placebo (N=30)
Muscle soreness (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No